CLINICAL TRIAL: NCT03546322
Title: Customized Registry Tool for Tracking Adherence to Clinical Guidelines for Head and Neck Cancers
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: P30HS023558-1; P30HS023558 (NIH)
Record Dates: First submitted 2018-05-10; First posted 2018-06-06 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Head and Neck Neoplasms
Keywords: head and neck cancer; health information technology; patient safety; adherence; ambulatory; outpatient; human factors; vulnerable populations; chronic disease
MeSH Terms: conditions — Head and Neck Neoplasms; Chronic Disease | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Registry: Head and neck cancer patients monitored on registry
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Patients who are diagnosed with head and neck cancer and monitored by the Otolaryngology - Head and Neck Surgery clinic at Zuckerberg San Francisco General Hospital and Trauma Center will be included in this group. The intervention is the implementation of a registry, designed to replace existing paper-based systems for tracking patients. All head and neck cancer patients monitored by the clinic will be included.

SUMMARY:
To implement and evaluate a health information technology platform designed to support the management of patients with head and neck cancer in an urban, publicly-funded outpatient setting. This is an observational study; researchers will not assign specific interventions to study participants.

DETAILED DESCRIPTION:
The investigators aim to implement and evaluate a health information technology (HIT) registry at an urban, public delivery system. The investigators will not assign specific interventions to the study participants, but rather observationally assess the effect of the HIT registry, designed to support routine medical care, on participants.

The investigators will use systems engineering methodologies to design, develop, and implement the platform. The platform will be implemented in the Otolaryngology - Head and Neck Surgery clinic that cares for patients with head and neck cancers. The study will assess patient outcomes and evaluate the time it takes for patients to progress through key treatment and post-treatment milestones before and after the HIT tool is implemented. The investigators will use models controlling for secular trend to estimate the effect of the tool on improving timely and successful completion of guideline-based care processes.

The HIT platform seeks to improve the monitoring and alerting functionality of existing systems. Specifically, it replaces paper-based systems previously used by the clinic to monitor its head and neck cancer patients. It will be implemented clinic-wide for all patients being treated for head and neck cancers. The investigators are not assigning a specific intervention to patients, but rather supporting the clinic and health system in the development of a population management platform that improves routine care processes. The platform is approved for clinical use and research by the San Francisco Health Network and the University of California, San Francisco.

The HIT platform users are clinicians who are responsible for monitoring patients with head and neck cancer and agree to partner with the investigators to improve monitoring processes. The clinicians involved may be asked to voluntarily participate in surveys, interviews, focus groups, and program evaluations. Patient medical records will be reviewed, but patients monitored on the registry will not be contacted by researchers.

Procedures are in place to monitor the registry. First, quality assurance is performed by the research team, information technology analysts, and software engineers. This includes checking that data in the platform matches source data, such as data entered in the electronic health record. In addition, the platform users are audited on a weekly basis. A data dictionary defining variables used in the platform exists and is updated as needed. Patients will be added to the registry by a clinician if they are diagnosed with head and neck cancer. The research team will support the clinicians in data analysis, although this will be performed with population-level, de-identified data. However, if unmediated adverse events are identified by the research team, the research team will alert the clinicians immediately. The HIT platform is designed to supplement, but not replace, the existing electronic health record. Data on the registry will be validated with source data and users will still engage with the source data and electronic health record as appropriate clinically and operationally.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck surgery monitored by the Otolaryngology - Head and Neck Surgery Clinic

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer monitored by the Otolaryngology - Head and Neck Surgery clinic at the Zuckerberg San Francisco General Hospital and Trauma Center
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Workup and Treatment Planning - Primary Outcome | From date of diagnosis to first date of treatment, assessed up to 5 years
  Time from diagnosis to initiation of treatment
Treatment - Primary Outcome | 5 years
  Proportion of patients that complete tumor board treatment recommendations

SECONDARY OUTCOMES:
Workup and Treatment Planning - Secondary Outcome #1 | From date of diagnosis to presentation at tumor board, assessed up to 5 years
  Time from diagnosis to presentation at tumor board
Workup and Treatment Planning - Secondary Outcome #2 | From date of diagnosis to date of dental evaluation for patients undergoing radiation treatment, assessed up to 5 years
  Time from diagnosis to dental evaluation
Workup and Treatment Planning - Secondary Outcome #3 | From date of diagnosis to date of first visit with oncology clinic, assessed up to 5 years
  Time from diagnosis to first visit in oncology clinics
Treatment - Secondary Outcome | 6 weeks
  Proportion of patients who complete post-treatment radiation
Loss to follow-up | 5 years
  Proportion of patients who are lost to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Urmimala Sarkar, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hickey MD, Lisker S, Brodie S, Vittinghoff E, Russell MD, Sarkar U. Customized registry tool for tracking adherence to clinical guidelines for head and neck cancers: protocol for a pilot study. Pilot Feasibility Stud. 2020 Feb 7;6:16. doi: 10.1186/s40814-020-0552-0. eCollection 2020. PMID 32047648